CLINICAL TRIAL: NCT06694389
Title: A Phase 3, Randomized, Observer-Blind, Active-Control Study to Evaluate the Immunogenicity, Reactogenicity, and Safety of mRNA-1083 (SARS-CoV-2 and Influenza) Vaccine in Healthy Adults ≥50 Years of Age
Brief Title: Study to Investigate the Immunogenicity, Reactogenicity, and Safety of mRNA-1083 Vaccine (SARS-CoV-2 [COVID-19] and Influenza) in Adults ≥50 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mRNA-1083-P302
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: COVID-19; Influenza
Keywords: Influenza; COVID-19; Messenger RNA; Moderna
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — COVID-19 Vaccines; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- mRNA-1083 and Placebo (Experimental): Participants 50 years of age and older will receive mRNA-1083 by intramuscular (IM) injection and placebo by subcutaneous (SC) or IM injection administered on Day 1.
  Interventions: Biological: mRNA-1083; Other: Placebo
- Licensed influenza vaccine + SARS-CoV-2 vaccine (Active Comparator): Participants of age 50 years and older will receive licensed influenza vaccine by SC or IM injection and SARS-CoV-2 vaccine by IM injection administered on Day 1.
  Interventions: Biological: Licensed Influenza Vaccine; Biological: SARS-CoV-2 Vaccine

INTERVENTIONS:
Biological: mRNA-1083 — Suspension for injection
  Arms: mRNA-1083 and Placebo
Other: Placebo — 0.9% sodium chloride suspension for injection
  Arms: mRNA-1083 and Placebo
Biological: Licensed Influenza Vaccine — Aqueous injectable (SC) or suspension for injection (IM)
  Other Names: Influenza HA, Biken, and; Fluarix tetra
  Arms: Licensed influenza vaccine + SARS-CoV-2 vaccine
Biological: SARS-CoV-2 Vaccine — Suspension for injection
  Other Names: mRNA-1273
  Arms: Licensed influenza vaccine + SARS-CoV-2 vaccine

SUMMARY:
The purpose of the study is to evaluate the immunogenicity, reactogenicity, and safety of mRNA-1083 in adults 50 years of age and older in participating countries (Japan, Taiwan, and South Korea).

ELIGIBILITY:
Key Inclusion Criteria:

* Medically stable adults ≥50 years of age at the time of consent (Screening/Day 1 Visit).
* A participant who could become pregnant is eligible to participate if the following is met:

  * Not pregnant or breast/chestfeeding, and is using a contraceptive method that is highly effective for at least 90 days after the study intervention administration and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period.
  * Have a negative highly sensitive pregnancy test (urine) as required by local regulations at Screening/Day 1 Visit, before the study intervention.
* Participants who can produce sperm are eligible to participate if they agree to the following for at least 90 days after the study intervention administration:

  * Refrain from donating sperm.
  * Either be abstinent from reproductive sexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use an external condom with a person who could become pregnant partner use of an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse.
* Agree to use an external condom when engaging in any activity that allows for passage of ejaculate to another person.
* Received ≥2 COVID-19 vaccines and the last COVID-19 vaccine was ≥150 days prior to Day 1

Key Exclusion Criteria:

* History of a diagnosis or condition that, in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of study endpoints, assessment of immune response, or adherence to study procedures.
* Any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Known history of SARS-CoV-2 infection within 150 days prior to Day 1.
* Tested positive for influenza by local health authority-approved testing methods ≤150 days prior to Day 1.
* Received corticosteroids at ≥10 mg/day of prednisone or equivalent for >14 days in total within 90 days prior to Day 1 or is anticipating the need for corticosteroids at any time during the study. Inhaled nasal and topical steroids are allowed.
* Received systemic immunosuppressive treatment, including long-acting biological therapies that affect immune responses (for example, infliximab), within 180 days prior to Day 1 or plans to do so during the study.
* Received or plans to receive any vaccine authorized or approved by a local health agency ≤28 days prior to study injections or plans to receive a vaccine authorized or approved by a local health agency within 28 days after the study injections.
* Received a seasonal influenza vaccine ≤150 days prior to Day 1.
* Treated with antiviral therapies for influenza (for example, Tamiflu®) ≤150 days prior to Day 1.
* Has had close contact with someone with laboratory-confirmed influenza infection or with someone who has been treated with antiviral therapies for influenza (for example, Tamiflu) within 5 days prior to Day 1
* Has had close contact to someone with COVID-19 as defined by the Centers for Disease Control and Prevention (CDC) in the past 10 days prior to Day 1.
* Has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit/Day 1 or plans to donate blood products during the study.
* Reported history of anaphylaxis or severe hypersensitivity reaction after receipt of any mRNA or influenza vaccines or any components of the mRNA or influenza vaccines, including egg protein.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2457 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Geometric Mean (GM) Level of Antibodies for Influenza, as Measured by Hemagglutination Inhibition (HAI) Assay | Day 29
GM Level of Antibodies for SARS-CoV-2, as Measured by Pseudovirus Neutralization Assay (PsVNA) | Day 29
Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) | Day 1 through 7 days after study injection
Number of Participants With Unsolicited Adverse Events (AEs) | Day 1 through 28 days after study injection
Number of Participants With Medically Attended Adverse Events (MAAEs) | Day 1 though Day 181
Number of Participants With Adverse Events of Special Interest (AESIs) | Day 1 though Day 181
Number of Participants With Serious Adverse Events (SAEs) | Day 1 through Day 181
Number of Participants With AEs Leading to Discontinuation | Day 1 through Day 181

SECONDARY OUTCOMES:
Influenza: Percentage of Participants with Seroconversion, as Measured by HAI Assay | Day 29
  Seroconversion is defined as a Day 29 post-injection level ≥1:40 if baseline is <1:10 or a 4-fold or greater rise if baseline is ≥1:10 in anti-HA antibodies measured by HAI assay.
SARS-CoV-2: Percentage of Participants with Seroresponse, as Measured by PsVNA | Day 29
  Seroresponse is defined as a Day 29 post-injection level ≥4-fold if baseline is ≥lower limit of quantification (LLOQ) or ≥4*LLOQ if baseline titer is <LLOQ in neutralizing antibody (nAb) values measured by PsVNA.
Geometric Mean Fold-Rise (GMFR) of Antibodies for Influenza, as Measured by HAI Assay | Day 1, Day 29
GMFR of Antibodies for SARS-CoV-2, as Measured by PsVNA | Day 1, Day 29

CONTACTS AND LOCATIONS:
Locations (44):
- Japan (26):
  - Public Health Association.Inc., Nagoya, Aichi-ken
  - Daido Clinic, Nagoya, Aichi-ken
  - Tenjin Sogo Clinic, Fukuoka, Fukuoka
  - PS Clinic - Internal medicine, Fukuoka, Fukuoka
  - Fukuoka Heartnet Hospital, Fukuoka, Fukuoka
  - Medical Coporation of Yamazaki Neurotology, Rhinolaryngology Clinical, Sapporo, Hokkaido
  - Motomachi Takatsuka Naika Clinic - Internal Medicine, Yokohama, Kanagawa
  - Sakurajyuji Medical Corporation Medimesse Sakurajyuji Clinic, Kumamoto, Kumamoto
  - Nishi-Kumamoto Hospital, Kumamoto, Kumamoto
  - Sato Hospital, Osaki-shi, Miyagi
  - Yokoi Medicine Clinic, Mino, Osaka
  - Shinwakai Adachi Kyosai Hospital - Internal Medicine, Adachi-ku, Tokyo
  - Dojinkinenkai Meiwa Hospital, Chiyoda-ku, Tokyo
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Tokyo center clinic - Internal medicine, Chuo-ku, Tokyo
  - Medical Corporation Asbo Tokyo Asbo Clinic, Chuo-ku, Tokyo
  - New Medical Research System Clinic, Hachioji-shi, Tokyo
  - Shimamura Memorial Hospital, Nerima City, Tokyo
  - Denenchofu Family Clinic, Ōta-ku, Tokyo
  - Hillside Clinic Jingumae, Shibuya-ku, Tokyo
  - Clinical Research Tokyo Hospital - Clinical Research Center, Shinjuku, Tokyo
  - Higashi-Shinjuku Clinic - Internal Medicine, Shinjuku, Tokyo
  - Shinei Medical Healthcare Clinic, Suginami, Tokyo
  - Souseikai Sumida Hospital, Sumida-Ku, Tokyo
  - Seishukai Clinic, Taito-ku, Tokyo
  - Metropolitan Clinic - Internal Medicine, Toshima-ku, Tokyo
- South Korea (10):
  - Korea University Ansan Hospital, Ansan-si
  - Kyungpook National University Hospital - Infectious Diseases, Daegu
  - Chonnam National University Hospital - Allergology, Gwangju
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju
- Taiwan (8):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kuang Tien General Hospital - Dajia, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital - Neihu Branch - Infectious Diseases, Taipei
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital, Taoyuan District